CLINICAL TRIAL: NCT01990677
Title: Eplerenone for the Treatment of Central Serous Chorioretinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Collaborators: Mid Atlantic Retina (Other)
Responsible Party: Principal Investigator, MidAtlantic Retina, Dr. Mitchell Fineman, Wills Eye
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: ECSelsior; ESCelsior2013 (Other: Mid Atlantic Retina)
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Results first posted 2017-06-29 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-10

CONDITIONS: Central Serous Chorioretinopathy
Keywords: Central Serous Chorioretinopathy; csr; cscr; eplerenone; vision; choroid; retina; acute; chronic
MeSH Terms: conditions — Central Serous Chorioretinopathy; Bronchiolitis Obliterans Syndrome | interventions — Eplerenone; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 25mg Eplerenone- Chronic CSCR Diagnosis (Active Comparator): Dosing will begin at 25mg Eplerenone taken orally , one time, each day for 58 days. Throughout the 58 day treatment period dosage will be adjusted. The adjustment will be based on serum potassium and creatine levels from blood draws done at Day 12 and Day 33. From the 25 mg starting dosage, the dosage will either be increased to 50 mg a day or reduced to placebo, one time, each day.
  Interventions: Drug: 25mg Eplerenone; Drug: Placebo
- Placebo- Chronic CSCR Diagnosis (Placebo Comparator): Dosing will begin with placebo and will stay as placebo throughout the study. The placebo pills will be taken orally, once daily, for 58 days. The placebo pills will be compounded to be of similar composition to the eplerenone tablets, without the active ingredient.
  Interventions: Drug: Placebo
- 25mg Eplerenone- Acute CSCR Diagnosis (Active Comparator): Dosing will begin at 25mg Eplerenone taken orally , one time, each day for 28 days. Throughout the 28 day treatment period, dosage will be adjusted based on serum potassium and creatine levels from blood draws done on Day 12. From the 25 mg starting dosage, the dosage will either be increased to 50 mg a day or reduced to placebo, one time, each day.
  Interventions: Drug: 25mg Eplerenone; Drug: Placebo
- Placebo- Acute CSCR Diagnosis. (Active Comparator): Dosing will begin with placebo and will stay as placebo throughout the study. The placebo pills will be taken orally, once daily, for 28 days. The placebo pills will be compounded to be of similar composition to the eplerenone tablets, without the active ingredient.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 25mg Eplerenone — Patients will be given 25mg Eplerenone (or 50mg Eplerenone) or placebo throughout the study and the dosage will be based on the serum potassium/creatine levels. Patients will be randomized 2:1 such that 36 patients in each group will receive eplerenone and 16 patients in each group will receive placebo
  Other Names: Eplerenone; Inspra
  Arms: 25mg Eplerenone- Acute CSCR Diagnosis; 25mg Eplerenone- Chronic CSCR Diagnosis
Drug: Placebo — Patients will be given placebo throughout the study from day one, other patients may be tapered down to placebo based on the serum potassium/creatine levels. 16 patients in each group will receive placebo.
  Other Names: Sugar pill

SUMMARY:
To test the effect oral eplerenone versus placebo in patients with central serious chorioretinopathy .

DETAILED DESCRIPTION:
To evaluate the effect of oral eplerenone compared to placebo in patients with central serous chorioretinopathy (CSCR) on sub-foveal (small part of retina) fluid using optical coherence tomography (OCT).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Ability to give written informed consent
* Sub-retinal fluid under fovea seen on OCT
* Diagnosis of central serous chorioretinopathy (CSCR): classification is at the discretion of the investigator, but general guidelines are

  1. Acute- first episode or symptoms less than one month prior to presentation
  2. Chronic- previously documented sub-foveal fluid, any prior treatment, symptoms for over 3 months, or <50% reduction in fluid thickness on OCT after 3 months.

Exclusion Criteria:

* Age under 18
* Impaired decision-making ability
* At initial laboratory screening serum potassium >5.5 milliequivalent (mEq)/L
* At initial laboratory screening serum creatinine >2 mg/dL in men and >1.8 mg/dL in women or decreased renal function by creatinine clearance less than 50 mL/min
* Absence of sub-foveal fluid
* Any patient with prior treatment for CSCR within 3 months of enrollment
* Patients taking potassium supplements or potassium-sparing diuretics spironolactone, amiloride, and triamterene and/or potent CYP3A4 (cytochrome) inhibitors (amifostine, cyclosporine, fluconazole, itraconazole, ketoconazole, mifepristone, posaconazole, potassium salts, rituximab, tacrolimus, voriconazole nefazodone, troleandomycin, clarithromycin, ritonavir, and nelfinavir)
* Women who are pregnant or are actively trying to conceive
* Patients with type 1 or type 2 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2013-10; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Fineman, MD, Principal Investigator — Mid Atlantic Retina
Locations (10):
- United States (10):
  - Mid Atlantic Retina, Cherry Hill, New Jersey
  - Mid Atlantic Retina, Marlton, New Jersey
  - Mid Atlantic Retina, Mays Landing, New Jersey
  - Mid Atlantic Retina, Bala-Cynwyd, Pennsylvania
  - Mid Atlantic Retina, Bethlehem, Pennsylvania
  - Mid Atlantic Retina, Huntingdon Valley, Pennsylvania
  - Mid Atlantic Retina, Lansdale, Pennsylvania
  - Mid Atlantic Retina, New Wilmington, Pennsylvania
  - Mid Atlantic Retina, Newtown Square, Pennsylvania
  - Mid Atlantic Retina, Plymouth Meeting, Pennsylvania

REFERENCES:
- [Derived] Lange CA, Qureshi R, Pauleikhoff L. Interventions for central serous chorioretinopathy: a network meta-analysis. Cochrane Database Syst Rev. 2025 Jun 16;6(6):CD011841. doi: 10.1002/14651858.CD011841.pub3. PMID 40522203

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Significant acute data collection missing therefore only chronic arm data analysis was reviewed and entered into results data.
Period: Overall Study
Arm/Group | 25mg Eplerenone- Chronic CSCR Diagnosis | Placebo- Chronic CSCR Diagnosis
Started | 12 | 6
Completed | 10 | 5
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Population: Two individuals in the treatment group and one in the placebo group were lost to follow-up.
Groups:
- Total: Total of all reporting groups
Arm/Group | 25mg Eplerenone- Chronic CSCR Diagnosis | Placebo- Chronic CSCR Diagnosis | Total
Number analyzed (Participants) | 10 | 5 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 4 | 13
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (11.8) | 62 (5.5) | 54 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 8 | 4 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Maximal Subretinal Fluid Height Based on Spectral Domain Optical Coherence Tomography (OCT) Measurement.
Description: Mean change in maximal subretinal fluid height based on spectral domain OCT from baseline to month 2 in chronic central serous chorioretinopathy (CSCR) patients receiving placebo versus eplerenone.
Time Frame: Baseline and 2 months
Population: Significant acute data collection missing therefore only chronic arm data analysis was reviewed and entered into results data.
Measure: Mean (Standard Deviation); unit: microns
Units Other Than Participants: Eyes
Arm/Group | 25mg Eplerenone- Chronic CSCR Diagnosis | Placebo- Chronic CSCR Diagnosis
Number analyzed (Participants) | 10 | 5
Number analyzed (Eyes) | 15 | 6
microns
  Baseline | 139.3 (58.7) | 135.9 (21.8)
  Month 2 | 51.8 (52.2) | 172.3 (88.8)

2. Secondary Outcome: Mean Change in Subfoveal Fluid Height Based on OCT Measurement
Description: Mean change in subfoveal fluid height based on spectral domain OCT measurement from baseline to month 2 in chronic CSCR patients receiving placebo versus eplerenone.
Time Frame: Baseline and Month 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microns
Units Other Than Participants: Eyes
Arm/Group | 25mg Eplerenone- Chronic CSCR Diagnosis | Placebo- Chronic CSCR Diagnosis
Number analyzed (Participants) | 10 | 5
Number analyzed (Eyes) | 15 | 6
microns
  Baseline | 121.4 (75.0) | 92.1 (47.4)
  Month 2 | 29.4 (34.0) | 134.0 (105.9)

3. Other Pre Specified Outcome: Proportion of Eyes Demonstrating a Reduction in Subretinal Fluid on OCT
Description: Proportion of eyes having a decrease in subretinal fluid on spectral domain OCT from baseline to month 2 in chronic CSCR patients receiving placebo versus eplerenone.
Time Frame: Baseline and Month 2
Population: as for outcome 1
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | 25mg Eplerenone- Chronic CSCR Diagnosis | Placebo- Chronic CSCR Diagnosis
Number analyzed (Participants) | 10 | 5
Number analyzed (Eyes) | 15 | 6
Eyes | 11 | 1

ADVERSE EVENTS:
Description: Significant acute data collection missing therefore only chronic arm data analysis was reviewed and entered into results data.
Arm/Group | 25mg Eplerenone- Chronic CSCR Diagnosis | Placebo- Chronic CSCR Diagnosis
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6
Other Adverse Events (participants affected / at risk) | 1/12 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 25mg Eplerenone- Chronic CSCR Diagnosis (N=12) | Placebo- Chronic CSCR Diagnosis (N=6)
Dizziness (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No